CLINICAL TRIAL: NCT06229600
Title: Respiratory Rehabilitation and the Impact of Psychiatric Comorbidities
Brief Title: REspiratory reHABilitation and PSYchiatric Comorbidities
Acronym: REHABPSY
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: CET 2023-3.11/439.1
Record Dates: First submitted 2023-12-29; First posted 2024-01-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Disease
Keywords: Chronic respiratory insufficiency; Cognitive impairment; Mental Health; COPD; Lung diseases
MeSH Terms: conditions — Respiration Disorders; Cognitive Dysfunction; Psychological Well-Being; Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group A: Patients with an established diagnosis according to the DSM-5 classification (DIAGNOSTIC AND STATISTICAL MANUAL OF MENTAL DISORDERS - FIFTH EDITION, 2014) and possible drug therapy (24).
  * Schizophrenia spectrum disorders and other psychotic disorders
  * Bipolar disorder and related disorders
  * Depressive disorders
  * Anxiety disorders
  * Obsessive-compulsive disorder and related disorders
  * Disorders related to traumatic and stressful events
  * Dissociative disorders
  * Somatic symptoms and related disorders
  * Nutrition and eating disorders
  * Evacuation disorders
  * Sleep-wake disorders
  * Sexual dysfunctions
  * Gender dysphoria
  * Disruptive behaviour, impulse control and conduct disorder
  * Substance-related and addiction disorders
  * Personality disorders
  * Paraphilia disorders
  * Autism spectrum disorders
  * ADHD
  Interventions: Other: Standard rehabilitation
- Group B: Patients on medication (psychotropic drugs) without a reported/reported specific psychiatric diagnosis in their clinical history.
  Interventions: Other: Standard rehabilitation
- Group C: Patients without a history/reported psychiatric disorder and without specific psychopharmacological therapy.
  Interventions: Other: Standard rehabilitation
- Group D: Patients with a history of diagnosed neurocognitive disorder.
  Interventions: Other: Standard rehabilitation
- Group E: Patients in the practice without a history/report of psychiatric disorders and without specific psychopharmacological treatment on admission who are diagnosed during admission.
  This is a subgroup of the C group.
  Interventions: Other: Standard rehabilitation
- Group F: Patients in the practice without a history/report of psychiatric disorders and without specific psychopharmacological therapy on admission who are diagnosed during admission for suspected psychiatric/neurocognitive pathology and are discharged with indications for further investigation at the territorial services.
  This is a subgroup of the C group.
  Interventions: Other: Standard rehabilitation

INTERVENTIONS:
Other: Standard rehabilitation — Respiratory rehabilitation

SUMMARY:
Patients with respiratory insufficiency, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, asthma, bronchiectasis, and, to a lesser extent, other pathologies that result in respiratory insufficiency and require rehabilitation are admitted to in-hospital Respiratory Rehabilitation. Several studies have assessed the impact of comorbidities in the most frequent respiratory diseases such as COPD, asthma, pulmonary fibrosis, and cystic fibrosis in terms of worsening mortality, morbidity, and disease progression.

However, to our knowledge, there is no reliable quantification in Italy of the percentage of the presence of mental disorders (psychiatric/neurodegenerative) according to the Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-5 classification in respiratory patients as well as the prevalence of mental disorders present among patients requiring in-hospital rehabilitation programs.

The study hypothesizes that these disorders are present among patients admitted to rehabilitation centers and that they may impact the final rehabilitation outcome.

DETAILED DESCRIPTION:
Patients with respiratory insufficiency, COPD, pulmonary fibrosis, asthma, bronchiectasis, and, to a lesser extent, other pathologies that result in respiratory insufficiency and require rehabilitation are admitted to in-hospital Respiratory Rehabilitation. Several studies have assessed the impact of comorbidities in the most frequent respiratory diseases such as COPD, asthma, pulmonary fibrosis, and cystic fibrosis in terms of worsening mortality, morbidity, and disease progression.

Comorbidities have been studied and assessed by scales such as the COTE, the Charlson comorbidity index (CCI), and the Cumulative Illness Rating Scale (CIRS). These comorbidities assessed predominantly focus on metabolic and cardiovascular aspects and only a small number of studies considered psychiatric comorbidity, mainly depression.

In previous studies depression, anxiety and psychiatric disease were 8th, 14th, and 23rd in frequency as comorbidity.

Other, more evaluated comorbidities were high blood pressure (17%-64.7%), coronary artery disease (19.9%-47.8%), diabetes mellitus (10.2%-45%) osteoarthritis (18%-43.8%), psychiatric conditions (12.1%-33%) and asthma (14.7%-32.5%).

Among psychological/psychiatric/neurodegenerative comorbidities, anxiety, and depression have been more extensively studied, with worse rehabilitation outcomes, more symptoms (especially dyspnoea), less functional exercise capacity, and minor quality of life (QOL). Similarly, patients with COPD and obstructive sleep apnea syndrome (OSAS), as demonstrated in numerous studies, are more frequently affected by neurocognitive disorders.

Gender differences in reporting psychiatric and respiratory comorbidity have been previously observed: twice as many psychiatric disorders in women as in men, and with higher levels of anxiety and depression in women than in men.

Pulmonary diseases are historically and etiologically related to smoking and unfavorable environmental exposures, two factors that are more present in less affluent social groups, where an increase in psychiatric diseases is known. People with psychiatric diseases and fewer contextual resources also arrive later to be diagnosed with COPD and/or lung cancer, thus leading to a more unfavorable course.

Respiratory rehabilitation is for some respiratory diseases the standard of care among non-pharmacological therapies and should possibly lead to a return to a state of health identified as the person's 'well-being'. As recently published in a study conducted by the Italian Health Ministry, only 18% of Italians feel in a state of full well-being, understood as a state of complete physical, mental, and social well-being and not simply the absence of disease', indicating how complex it is to achieve this state, particularly for people with respiratory pathologies.

In recent years, therefore, there has been growing scientific evidence that there is a close correlation between mental and physical health to achieve maximum well-being also understood as 'the ability to adapt and self-manage in the face of social, physical and emotional challenges. For some years now, and even more after the recent severe acute respiratory syndrome (SARS)-CoV-2 pandemic outbreak, more and more attention has been paid to psychological and psychiatric disorders, especially anxiety, depression, and substance abuse.

Patients admitted to in-hospital respiratory rehabilitation often have complex comorbidities that affect recovery after an acute event.

These studies suggest that psychiatric/neurodegenerative pathologies may therefore significantly impact the patient's condition by increasing the risk of developing pulmonary disease, slowing down diagnosis and treatment, and acting as a brake on the possibility of deriving maximum benefit from pharmacological and non-pharmacological treatments such as rehabilitation and the continuation of adequate chronic disease management at home.

To our knowledge, there is no reliable quantification in Italy of the percentage of the presence of mental disorders (psychiatric/neurodegenerative) according to the DSM-5 classification in respiratory patients as well as the prevalence of mental disorders present among patients requiring in-hospital rehabilitation treatment.

The study hypothesizes that these disorders are present among patients admitted to rehabilitation centers and that they may impact the final rehabilitation outcome for various reasons, including a reduced awareness of one's health condition, greater difficulty in therapeutic adherence, the ability to self-monitor, the reduction of risk factors and a reduced availability of resources. This also results in reduced effectiveness of the education provided.

The presence of mental disorders also has a significant impact on family members and caregivers who should ultimately participate in the full implementation of the rehabilitation project. We consider as important to evaluate this aspect as well with this Italian-based survey.

With this study we therefore intend to assess in our Institutes how many people arrive with a diagnosis and/or treatment for mental disorders, how many need attention, and how many are identified or suspected to be affected by a psychiatric/neurodegenerative disease during their stay, during routine assessments, collecting clinical history, treatment and comorbidities. Treating the patient as a clinical team with multiple approaches, it can be argued that clinically significant signs and symptoms of psychiatric/neurocognitive disorders are detected with adequate accuracy even in the absence of formal psychiatric assessment, which would make the study unduly burdensome in the setting of interest and could undermine patient acceptance.

All adult patients consecutively admitted for a course of Respiratory Rehabilitation - in 12 months - to the Units of Respiratory Rehabilitation belonging to the Department of Pneumology of the Maugeri Scientific Clinical Institutes will be studied. On admission (T0), anthropometric, clinical history (comorbidities measured with CIRS scale, presence of chronic respiratory failure (CRF), oxygen (O2) use, smoking history with number of packs/year, drug therapy, number of respiratory flare-ups per year, number of respiratory hospitalizations per year, days since respiratory index event, admission diagnosis, and current medication history will be collected.

Moreover:

* Frailty assessment: Sunfrail tool (ST) is a questionnaire for measuring frailty among older people. ST is a 9-item questionnaire consisting of nine questions selected from evidence-based tools already used in health services in the European Union and the USA to identify frailty in the bio (physical), psycho (cognitive and psychological), and social domains. The answer can be yes or no. Important is the percentage of yes, and important is frailty.
* Pulmonary function assessment of forced expiratory volume at one second (FEV1), forced vital capacity (FVC), and FEV1/FVC; if the patient is respiratory insufficient: saturation of oxygen (SatO2) in oxygen/air, oxygen desaturation index (ODI)/h, average night SatO2, and time under 90% oxygen saturation (T<90).
* Psychological/neuropsychological assessment by the Centre's psychologists only if specifically requested during the rehabilitation program by the relevant clinician.
* Sleep survey: Insomnia Severity Index. Designed as a brief screening tool for insomnia, the seven-item questionnaire Insomnia Severity Index (ISI) asks respondents to rate the nature and symptoms of their sleep problems using a Likert-type to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).

At the time of discharge from rehabilitation, patients will be classified according to the group A-F definition.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age, of either sex, eligible for admission to a Respiratory Rehabilitation Unit and who have signed the informed consent attesting to the patient's voluntary participation.

Exclusion Criteria:

* Patients unable to read, with significant speech and hearing impairment,or refusing participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: On admission (T0), clinical history, admission diagnosis, and current medication history will be collected for all patients admitted for respiratory rehabilitation. All patients will follow their tailored rehabilitation program according to the medical indication. At the time of discharge, they will be classified into six groups (A-F) according to the presence/absence of a psychiatric/cognitive diagnosis and/or pharmacological therapy.
Sampling Method: Non-Probability Sample
Enrollment: 994 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency of patients with or without comorbidities of psychiatric/neurocognitive disorders present on discharge from a respiratory rehabilitation program | At one month
  To quantify the percentage of patients in the study with or without comorbidities of psychiatric/neurocognitive disorders present on discharge from a respiratory rehabilitation pathway as follows:
  1. established psychiatric diagnosis and drug therapy
  2. drug therapy (psychotropic drugs) without a specific psychiatric diagnosis reported/reported in the history
  3. no history/reported psychiatric disorder and no specific psychopharmacological therapy
  4. history of diagnosis of neurocognitive disorder
  5. absence of history/report of psychiatric disorders and without specific psychopharmacological treatment in inpatients receiving a diagnosis during admission
  6. absence of history/report of psychiatric disorders and without specific psychopharmacological therapy on admission who receive a diagnosis during admission for suspected psychiatric/neurocognitive pathology and are discharged with indications for further investigation at the territorial services

SECONDARY OUTCOMES:
Gender difference | At one month
  To assess whether there are differences in the presence of mental disorders between males and females and whether there are pathological pictures with different prevalence between men and women
Response to rehabilitation on disease impact: CAT | At baseline and one month
  To assess whether the different groups of patients present a different pattern of response to rehabilitation in terms of rehabilitation outcome, several tests will be performed both at admission and discharge:
  For disease impact, CAT will be used. CAT is a questionnaire that can help you and a doctor discuss the impact COPD has on your daily life.
  CAT asks questions about eight areas, prompting you to assign a score ranging from 0 to 5 for each area.
  A score of 0 means there's no impairment in that area. A score of 5 means severe impairment. Your overall score will range from 0 to 40. Higher scores indicate your COPD has a greater impact on your overall health and well-being.
Response to rehabilitation on motor disability: Barthel Index | At baseline and one month
  For motor disability, Barthel Index will be used both at admission and discharge. Barthel Index for Activities of Daily Living is an ordinal scale that measures a person's ability to complete activities of daily living (ADL).
  The Barthel Index measures the degree of assistance required by an individual on ten mobility and self-care ADL items. The ten items are scored with several points, and then a final score (maximum 100) is calculated by summing the points awarded to each functional skill. This allows the examiner to measure a patient's functional disability by quantifying their performance. The higher the score (100), the more independent the patient is in completing the measured ADLs. Higher scores also indicate the patient is more likely to return home, with varying degrees of assistance, following hospital discharge. The lower the score (0), the more dependent the patient is on ADL completion, and the more skilled care will be required at discharge.
Response to rehabilitation on frailty: BRASS | At baseline and one month
  For frailty assessment, BRASS will be used both at admission and discharge. BRASS was developed as part of a system of planning for total (non-relapsing) discharge, above all for patients over the age of 65. It facilitates the identification of those at risk of prolonged hospitalization and/or a complicated discharge procedure.
  According to the BRASS score, three risk classes will be identified by the nurse:
  1. low risk (score from 0 to 10): subjects that do not require special efforts for the organization of their resignation, disability is very limited;
  2. medium risk (score 11 to 19): patients with problems related to complex clinical situations that require discharge planning, but probably no risk of institutionalization;
  3. high risk (score greater than or equal to 20): subjects who reported problems and require a continuity of care, probably, in rehabilitation facilities or institutions.
Response to rehabilitation on dyspnea symptoms: Medical Research Council (MRC) | At baseline and one month
  For dyspnea symptoms, MRC will be used both at admission and discharge. This scale measures perceived respiratory disability, using the World Health Organization (WHO) definition of disability being "any restriction or lack of ability to perform an activity in the manner or within the range considered normal for a human being". The mMRC (Modified Medical Research Council) Dyspnoea Scale is used to assess the degree of baseline functional disability due to dyspnoea. It is useful in characterizing baseline dyspnoea in patients with respiratory diseases such as COPD. The mMRC breathlessness scale ranges from grade 0 to 4, where 4 is the worse score.
Response to rehabilitation on dyspnea symptoms: Barthel Dyspnoea Index (Bld) | At baseline and one month
  For dyspnea symptoms related to activities of daily living, Barthel Dyspnoea Index (Bld) will be used both at admission and discharge. BId is a recent dyspnea scale integrating ten daily life activities of the Barthel index and five categories of dyspnea sensation intensity. BId scale was reported to be reliable, sensitive, and adequate as a tool for measuring the level of dyspnea while performing daily life activities and the responsiveness after treatment. The total BId score ranges from 0 (no dyspnea) to 100 (maximum level of dyspnea). A decrease in BId score represents an improvement, whereas an increase in the score represents a worsening in symptoms.
Response to rehabilitation on effort tolerance: 6-Minute Walking Test (6MWT) | At baseline and one month
  For effort tolerance assessment, the 6-minute walking test (6MWT) will be used both at admission and discharge. The object of this test is to walk as far as possible for 6 minutes. The patient will walk back and forth along this course (demonstrate one lap) for six minutes. The patient may slow down if necessary. If the patient stops, I want you to continue to walk again as soon as possible. It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It is measured in meters, more meters best performance.
Prevalence of the anamnestic factors in all groups | At baseline
  To assess the prevalence of all anamnestic factors collected at admission in the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Principal Investigator — Istituti Clinici Scientifici Maugeri
Locations (6):
- Italy (6):
  - Istituti Clinici Scientifici Maugeri, Telese Terme, Benevento
  - Istituti Clinici Scientifici Maugeri, Lumezzane, Brescia
  - Istituti Clinici Scientifici Maugeri, Montescano, Pavia
  - Istituti Clinici Scientifici Maugeri, Bari
  - Istituti Clinici Scientifici Maugeri, Milan
  - Istituti Clinici Scientifici Maugeri, Pavia

IPD SHARING:
Plan to Share IPD: No
All collaborating centers will manage pseudo-anonymized data by a proper eCRF to the coordinating center (ICSM Lumezzane) at the end of each month for 12 months. Data will be collected in a unique database managed by a health professional external to the research.

REFERENCES:
- [Background] De Luca V, Femminella GD, Leonardini L, Patumi L, Palummeri E, Roba I, Aronni W, Toccoli S, Sforzin S, Denisi F, Basso AM, Ruatta M, Obbia P, Rizzo A, Borgioli M, Eccher C, Farina R, Conforti D, Mercurio L, Salvatore E, Gentile M, Bocchino M, Sanduzzi Zamparelli A, Viceconte G, Gentile I, Ruosi C, Ferrara N, Fabbrocini G, Colao A, Triassi M, Iaccarino G, Liotta G, Illario M. Digital Health Service for Identification of Frailty Risk Factors in Community-Dwelling Older Adults: The SUNFRAIL+ Study Protocol. Int J Environ Res Public Health. 2023 Feb 21;20(5):3861. doi: 10.3390/ijerph20053861. PMID 36900872
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Vitacca M, Paneroni M, Baiardi P, De Carolis V, Zampogna E, Belli S, Carone M, Spanevello A, Balbi B, Bertolotti G. Development of a Barthel Index based on dyspnea for patients with respiratory diseases. Int J Chron Obstruct Pulmon Dis. 2016 Jun 7;11:1199-206. doi: 10.2147/COPD.S104376. eCollection 2016. PMID 27354778
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Blaylock A, Cason CL. Discharge planning predicting patients' needs. J Gerontol Nurs. 1992 Jul;18(7):5-10. doi: 10.3928/0098-9134-19920701-05. PMID 1629535
- [Background] J. E. Cotes, D. J. Chinn, MRC questionnaire (MRCQ) on respiratory symptoms. Occupational Medicine 2007; 57 (5): 388. https://doi.org/10.1093/occmed/kqm051.